CLINICAL TRIAL: NCT03462914
Title: Comparative Study Between Different Approaches to CPA -Petroclival Meningiomas
Brief Title: Comparative Study Between Different Approaches to CPA-petroclival Meningiomas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shady abdel raheem hassan, principal investigator, Assiut University
Other Study IDs: CPA-petroclival meningiomas
Record Dates: First submitted 2018-03-01; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
• Give an effective treatment for CPA-petroclival meningiomas and can detect the best approach for these tumors.

. Improve the outcome of these patients and decease rate of recurrence.

DETAILED DESCRIPTION:
There are several lesions arising in the petroclival region. The most frequent tumor is the petroclival meningioma, followed by chondrosarcomas, chordomas, schwannomas of the cranial nerves V and VII, and other malignant tumors [1, 2, 3, 4, 5].

Petroclival meningiomas are tumors of the skull base that present a formidable challenge to surgical resection because of their deep location and relationship to vital neurovascular structures. In the majority of the cases they are benign tumors, but may involve or infiltrate the skull base bone, the dura mater, the brainstem, and all important neurovascular structures of this region. The petroclival region comprises the anatomical location of the body of the sphenoid bone, the anterior central portion of the occipital bone, and is bordered on the lateral aspect by the petrous apex. The roof of this space is formed by the petroclival ligaments and the tentorium. This space contains important neurovascular structures that are frequently involved or displaced by the tumor in a variable pattern. The basilar artery with its branches may be embedded or displaced by the meningioma. The petrosal vein is often displaced posteriorly by the tumor. Cranial nerves III and IV are usually displaced upwardly and the nerve VI is often surrounded by tumor. Petroclival meningiomas have their origin medial to cranial nerves V, VII, VIII, IX, X, and XI, and reach the tentorium . They frequently extend to the middle cranial fossa, cavernous sinus, prepontine space, and down to the foramen magnum. These tumors frequently compress the brainstem making total removal very difficult or impossible without neurologic deficits. cerebellopontine angle (CPA) and low clivus meningiomas may reach these areas. These lesions usually need different surgical approaches as transpetrosal approach ( anterior, modified and combined ) and retrosigmoid approach

ELIGIBILITY:
Inclusion Criteria:

* Patient with a single lesion .
* Patient with a denovo lesion.

Exclusion Criteria:

* Patient with recurrent lesions.
* Patient with lesions after adjuvant therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with meningioma
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
The success rate of surgery | 1 year
  complete resection of the tumor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spetzler RF, Hamilton MG, Daspit CP. Petroclival lesions. Clin Neurosurg. 1994;41:62-82. No abstract available. PMID 7842625